CLINICAL TRIAL: NCT00855270
Title: The Efficacy of a Single Dose IV Hydrocortisone Given Within 6 Hours of Exposure to a Traumatic Event in PTSD Prevention
Brief Title: Efficacy of Single Dose IV Hydrocortisone in Post Traumatic Stress Disorder (PTSD) Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SHEBA-09-6884-JZ-CTIL
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline (Placebo Comparator): An IV injection of saline will be administered to the control group in a double blind, randomized manner.
  Interventions: Drug: Placebo
- Hydrocortisone (Experimental): IV hydrocortisone will be given in a double blind random manner as the active treatment group
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Placebo — IV saline will be used as placebo for control
  Arms: saline
Drug: Hydrocortisone — A single dose 90-150mg of Intra Venous Hydrocortisone. 90mg will be administrated to participants weighing 45-59kg. 100mg will be administrated to participants weighing 60-69kg. 120mg will be administrated to participants weighing 70-89kg. 140mg will be administrated to participants weighing 90-99kg. 150mg will be administrated to participants weighing 100-120kg.
  Other Names: Hcort
  Arms: Hydrocortisone

SUMMARY:
This study is designed to test the hypothesis that a single Hydrocortisone intra venous injection within 6 hours post-trauma facilitates physiological recovery thereby preventing the development of Post Traumatic Stress Disorder (PTSD) in the months following the event. In the absence of such treatment (i.e., under placebo conditions), we hypothesize that a greater proportion of persons would develop PTSD (i.e., fail to recover from acute effects).

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled trial in which trauma victims are randomized to receive a single intravenous injection of either Hydrocortisone (90-150mg)or placebo within the first six hours following trauma exposure. To provide a pre-treatment baseline, participants will receive a medical and psychological evaluation prior to treatment. After two weeks the research assistant or study psychiatrist will perform behavioral ratings and complete history details pertaining to PTSD risk factors. Participants will be assessed again by the study psychiatrist or research assistants at 1, 3, 8 & 13 months. Eligible subjects will include men and women over the age of 21, who have been exposed to an event meeting the DSM-IV "A.1" criterion for trauma exposure, and who provide written, informed consent to participate in the study. In order to recruit persons who are more likely to be at risk for the development of PTSD, we will only randomize persons expressing marked anxiety, emotional distress or dissociation, as assessed by the Visual Analog Scales. Potential participants will be recruited from trauma victims arriving at the Chaim Sheba Medical Center Emergency Room.

ELIGIBILITY:
Inclusion Criteria:

1. Persons over the age of 21, who have been exposed to an event meeting the DSM-IV "A.1" criterion for trauma exposure, expressing marked anxiety, and/ or emotional distress and/or dissociation, as assessed by the Visual Analog Scales
2. Who provide written, informed consent to participate in the study.

Exclusion Criteria:

1. Physical injury that would contraindicate participation or interfere with a subject's ability to give informed consent or cooperate with the screening or collection of initial measures. Examples include severe burn injury, life-threatening medical or surgical condition, condition requiring surgical intervention under general anesthesia, as indicated by Abbreviated Injury Scale (AIS), or by clinical judgment;
2. Head injury involving confusion, loss of consciousness, or amnesia;
3. Medical conditions such as extreme obesity, psoriasis, herpes, Cushing's syndrome, current infectious disease, current viral disease, tuberculosis, unstable diabetes or hypertension, myasthenia gravis, and heart failure. Persons taking medications that can interfere with the HPA axis (e.g.,steroids, betablockers,indomethacin) will be excluded;
4. Weight below 45 or above 120 kg.
5. Pregnancy (in suggestive cases, a pregnancy test will be performed);
6. Traumatic exposure that reflects ongoing victimization (e.g., domestic violence) to which the subject is likely to be re-exposed during the study period.
7. Overt psychopathology, intoxication, or under the influence of substances.
8. Evidence or history of schizophrenia, bipolar, other psychotic condition;
9. Prior history of PTSD;
10. Current or past history of dementia, amnesia, or other cognitive disorder predating trauma exposure;
11. Assessed serious suicide risk.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is symptom severity at the end of the trial .This will be determined using the Clinician Administered PTSD Scale (CAPS), a scale with established reliability and good psychometric properties. | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Zohar, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Yehuda R, McFarlane AC, Shalev AY. Predicting the development of posttraumatic stress disorder from the acute response to a traumatic event. Biol Psychiatry. 1998 Dec 15;44(12):1305-13. doi: 10.1016/s0006-3223(98)00276-5. PMID 9861473
- [Background] Delahanty DL, Raimonde AJ, Spoonster E. Initial posttraumatic urinary cortisol levels predict subsequent PTSD symptoms in motor vehicle accident victims. Biol Psychiatry. 2000 Nov 1;48(9):940-7. doi: 10.1016/s0006-3223(00)00896-9. PMID 11074232
- [Background] Yehuda R, Yang RK, Buchsbaum MS, Golier JA. Alterations in cortisol negative feedback inhibition as examined using the ACTH response to cortisol administration in PTSD. Psychoneuroendocrinology. 2006 May;31(4):447-51. doi: 10.1016/j.psyneuen.2005.10.007. Epub 2005 Dec 20. PMID 16364555
- [Background] Yehuda R, Brand SR, Golier JA, Yang RK. Clinical correlates of DHEA associated with post-traumatic stress disorder. Acta Psychiatr Scand. 2006 Sep;114(3):187-93. doi: 10.1111/j.1600-0447.2006.00801.x. PMID 16889589
- [Background] Morgan CA 3rd, Southwick S, Hazlett G, Rasmusson A, Hoyt G, Zimolo Z, Charney D. Relationships among plasma dehydroepiandrosterone sulfate and cortisol levels, symptoms of dissociation, and objective performance in humans exposed to acute stress. Arch Gen Psychiatry. 2004 Aug;61(8):819-25. doi: 10.1001/archpsyc.61.8.819. PMID 15289280
- [Background] Delahanty DL, Raimonde AJ, Spoonster E, Cullado M. Injury severity, prior trauma history, urinary cortisol levels, and acute PTSD in motor vehicle accident victims. J Anxiety Disord. 2003;17(2):149-64. doi: 10.1016/s0887-6185(02)00185-8. PMID 12614659
- [Background] Charney DS, Deutch AY, Krystal JH, Southwick SM, Davis M. Psychobiologic mechanisms of posttraumatic stress disorder. Arch Gen Psychiatry. 1993 Apr;50(4):295-305. doi: 10.1001/archpsyc.1993.01820160064008. No abstract available. PMID 8466391
- [Background] Schelling G, Briegel J, Roozendaal B, Stoll C, Rothenhausler HB, Kapfhammer HP. The effect of stress doses of hydrocortisone during septic shock on posttraumatic stress disorder in survivors. Biol Psychiatry. 2001 Dec 15;50(12):978-85. doi: 10.1016/s0006-3223(01)01270-7. PMID 11750894
- [Background] Schelling G. Effects of stress hormones on traumatic memory formation and the development of posttraumatic stress disorder in critically ill patients. Neurobiol Learn Mem. 2002 Nov;78(3):596-609. doi: 10.1006/nlme.2002.4083. PMID 12559838
- [Background] Schelling G, Kilger E, Roozendaal B, de Quervain DJ, Briegel J, Dagge A, Rothenhausler HB, Krauseneck T, Nollert G, Kapfhammer HP. Stress doses of hydrocortisone, traumatic memories, and symptoms of posttraumatic stress disorder in patients after cardiac surgery: a randomized study. Biol Psychiatry. 2004 Mar 15;55(6):627-33. doi: 10.1016/j.biopsych.2003.09.014. PMID 15013832
- [Background] Schelling G, Roozendaal B, Krauseneck T, Schmoelz M, DE Quervain D, Briegel J. Efficacy of hydrocortisone in preventing posttraumatic stress disorder following critical illness and major surgery. Ann N Y Acad Sci. 2006 Jul;1071:46-53. doi: 10.1196/annals.1364.005. PMID 16891561
- [Background] Lupien SJ, Maheu F, Tu M, Fiocco A, Schramek TE. The effects of stress and stress hormones on human cognition: Implications for the field of brain and cognition. Brain Cogn. 2007 Dec;65(3):209-37. doi: 10.1016/j.bandc.2007.02.007. Epub 2007 Apr 26. PMID 17466428
- [Background] Harvey BH, Brand L, Jeeva Z, Stein DJ. Cortical/hippocampal monoamines, HPA-axis changes and aversive behavior following stress and restress in an animal model of post-traumatic stress disorder. Physiol Behav. 2006 May 30;87(5):881-90. doi: 10.1016/j.physbeh.2006.01.033. Epub 2006 Mar 6. PMID 16546226
- [Background] Cohen H, Zohar J, Gidron Y, Matar MA, Belkind D, Loewenthal U, Kozlovsky N, Kaplan Z. Blunted HPA axis response to stress influences susceptibility to posttraumatic stress response in rats. Biol Psychiatry. 2006 Jun 15;59(12):1208-18. doi: 10.1016/j.biopsych.2005.12.003. Epub 2006 Feb 3. PMID 16458266
- [Background] Cohen H, Zohar J. An animal model of posttraumatic stress disorder: the use of cut-off behavioral criteria. Ann N Y Acad Sci. 2004 Dec;1032:167-78. doi: 10.1196/annals.1314.014. PMID 15677404
- [Background] Cohen H, Matar MA, Buskila D, Kaplan Z, Zohar J. Early post-stressor intervention with high-dose corticosterone attenuates posttraumatic stress response in an animal model of posttraumatic stress disorder. Biol Psychiatry. 2008 Oct 15;64(8):708-717. doi: 10.1016/j.biopsych.2008.05.025. Epub 2008 Jul 17. PMID 18635156
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Carmi L, Zohar J, Juven-Wetzler A, Desarnaud F, Makotkine L, Bierer LM, Cohen H, Yehuda R. Promoter methylation of the glucocorticoid receptor following trauma may be associated with subsequent development of PTSD. World J Biol Psychiatry. 2023 Sep-Oct;24(7):578-586. doi: 10.1080/15622975.2023.2177342. Epub 2023 Mar 13. PMID 36748398
- [Derived] Carmi L, Zohar J, Weissman T, Juven-Wetzler A, Bierer L, Yehuda R, Cohen H. Hydrocortisone in the emergency department: a prospective, double-blind, randomized, controlled posttraumatic stress disorder study. Hydrocortisone during golden hours. CNS Spectr. 2023 Aug;28(4):457-463. doi: 10.1017/S1092852922000852. Epub 2022 Jun 9. PMID 35678177
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873
- [Derived] Zohar J, Yahalom H, Kozlovsky N, Cwikel-Hamzany S, Matar MA, Kaplan Z, Yehuda R, Cohen H. High dose hydrocortisone immediately after trauma may alter the trajectory of PTSD: interplay between clinical and animal studies. Eur Neuropsychopharmacol. 2011 Nov;21(11):796-809. doi: 10.1016/j.euroneuro.2011.06.001. Epub 2011 Jul 8. PMID 21741804